CLINICAL TRIAL: NCT03566433
Title: Early Postoperative Pain After Totally Extraperitoneal Endoscopic Technique (TEP) vs. Lichtenstein Hernioplasty in Inguinal Hernia Repair: a Prospective Randomized Multi-center Study
Brief Title: Postoperative Pain After Endoscopic TEP vs. Lichtenstein Hernioplasty in Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: Helsinki University Central Hospital (Other); North Karelia Central Hospital (Other); Mikkeli Central Hospital (Other); Päijänne Tavastia Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KuopioUH
Record Dates: First submitted 2018-06-12; First posted 2018-06-25 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Inguinal Hernia; Hernia
MeSH Terms: conditions — Hernia, Inguinal; Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic TEP surgery (Active Comparator): Routine total extraperitoneal technique surgery for inguinal hernia
  Interventions: Procedure: Tep surgery for inguinal hernia
- Open Lichtenstein hernioplasty (Active Comparator): Routine lichtenstein surgery for inguinal hernia
  Interventions: Procedure: Lichtenstein

INTERVENTIONS:
Procedure: Tep surgery for inguinal hernia — TEP surgery
  Arms: Endoscopic TEP surgery
Procedure: Lichtenstein — Lichtenstein surgery for inguinal hernia
  Arms: Open Lichtenstein hernioplasty

SUMMARY:
Immediate pain reaction and return to work after TEP or Lichtenstein hernia repair have not been studied. In this multicenter trial the patients are allocated to surgery using TEP (n=50) or Lichtenstein (n=50) technique. Pain and return to work are recorded postoperatively up to one month. Immediate and late complications are also analyzed.

DETAILED DESCRIPTION:
Patient characteristics are recorded before surgery. The adult patients with inguinal hernia are randomized into endoscopic totally extraperitoneal hernioplasty (TEP) or open Lichtenstein hernioplasty. Pain reaction to surgery and return to work are asked many times using questionnaire and pain diary (pain scores from 1h to 30 days after surgery). Surgical complications and use of pain killers are carefully recorded. Clinical examination is performed if necessary.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of symptomatic inguinal hernia Age 18-80

Exclusion Criteria:

Large scrotal hernia Bilateral hernia Symptom-free hernia Inguinal pain without clinical evidence of hernia Asa class≥3

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Pain scores (0-100) after surgery | from day 1 to 1 month postoperatively
  Patients report pain after the operation at rest, during exercise and coughing. Higher scores means worse outcome

SECONDARY OUTCOMES:
Number of operative complications | from day 1 to 1 month postoperatively
  Any minor or major complication
Number of re-operations | 1 month after the operation
  Any re-operation

CONTACTS AND LOCATIONS:
Overall Officials: Hannu Paajanen, Prof, Study Director — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Matikainen M, Vironen JH, Silvasti S, Ilves I, Kossi J, Kivivuori A, Paajanen H. A randomized clinical trial comparing early patient-reported pain after open anterior mesh repair versus totally extraperitoneal repair of inguinal hernia. Br J Surg. 2021 Dec 1;108(12):1433-1437. doi: 10.1093/bjs/znab354. PMID 34791044